CLINICAL TRIAL: NCT01468038
Title: Sentra PM (a Medical Food) and Trazadone in the Management of Sleep Disorders
Brief Title: A Double-blind Placebo Controlled Trial of Sentra PM, a Medical Food
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SentraPM102
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active trazodone and placebo (Active Comparator): trazodone 50mg with Sentra PM-like placebo
  Interventions: Drug: Trazodone
- placebo and active Sentra PM (Active Comparator): Trazodone-like placebo and Sentra PM
  Interventions: Other: Sentra PM
- Sentra PM and trazodone (Active Comparator): Active Sentra PM and active trazodone
  Interventions: Drug: Sentra PM and Trazodone (CoPack Kit Trazamine)
- placebo trazodone and placebo Sentra PM (Placebo Comparator): trazadone-like placebo and Sentra PM-like placebo
  Interventions: Drug: Placebo trazodone and placebo Sentra PM

INTERVENTIONS:
Drug: Trazodone — active trazodone and sentra pm-like placebo
  Arms: Active trazodone and placebo
Other: Sentra PM — Active Sentra PM and trazodone-like placebo
  Arms: placebo and active Sentra PM
Drug: Sentra PM and Trazodone (CoPack Kit Trazamine) — A CoPack Kit - Trazamine, consisting of the co-administration of Sentra PM and trazodone.
  Arms: Sentra PM and trazodone
Drug: Placebo trazodone and placebo Sentra PM — Trazodone-like placebo and Sentra PM-like placebo co-administered as placebo of Trazamine CoPack Kit.
  Arms: placebo trazodone and placebo Sentra PM

SUMMARY:
This is a double blind placebo controlled study of one hundred and four subjects which will be randomized for treatment with Sentra PM alone, Sentra PM with trazadone, trazadone alone and placebo alone. Twenty -six subjects will be randomly placed in one of the four groups. Each of the one hundred and four subjects will undergo baseline examination to include a sleep study questionnaires and 24- hour electrocardiographic recording. The one hundred and four subjects will then be randomly placed in one of the four groups.

DETAILED DESCRIPTION:
Sentra PM can induce restorative sleep compared to placebo, and as good as a sleep drug (trazadone) in subjects experiencing non-restorative sleep. Sentra PM taken with trazadone works better than either product alone. Twenty-six subjects will be randomized to a two week ingestion of Sentra PM at bedtime, twenty-six subjects will be randomized to a two week ingestion of trazadone at bedtime, twenty-six subjects will be randomized to a two week ingestion of Sentra PM with trazadone at bedtime and twenty -six subjects will be randomized to a two week ingestion of placebo at bedtime. Each morning after ingestion of either active product or placebo, the subject will fill out sleep questionnaires. On the fourteenth day of ingestion, a repeat 24-Hour ECG examination will be performed on all one hundred and four subjects and each subject will give a second blood sample for analysis. On the morning of the 14th day of ingestion the final sleep questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 and below age 65.
* Patients with a history of a sleep disturbance with non-restorative sleep defined by perceived increase in sleep latency or morning/daytime grogginess.

Exclusion Criteria:

* Subjects who have previously taken GABAdone, SentraPM or trazadone.
* Subjects who are currently taking tricyclic anti-depressants.
* Any blood chemistry anomalies the investigator finds that may put the patient at risk or invalidate study results.
* Pregnant or lactating females.
* Subjects with implanted pacemakers or other implanted electrical devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Time to fall asleep | 14 days
  Subjects time to fall asleep will be measure by patient response to questionnaires to determine if time improved, stayed the same or worsen.

SECONDARY OUTCOMES:
Quality of Sleep | 14 days
Morning grogginess | 14 days
Feelings of depression | 14 days
Feelings of anxiety | 14 days
Improvement in parasympathetic activity | 14 days
  Improved parasympathetic activity measured by 24 hour ECG holter moniter.

CONTACTS AND LOCATIONS:
Locations (1):
- Targeted Medical Pharma, Los Angeles, California, United States